CLINICAL TRIAL: NCT00816803
Title: Autologous Bone Marrow Derived Cell Transplant in Spinal Cord Injury Patients
Brief Title: Cell Transplant in Spinal Cord Injury Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Al-Azhar University (Other); Medical Military Academy, Egypt (Unknown); Alexandria University (Other)
Responsible Party: Hatem E. Sabaawy, M, PhD, Assistant Professor of Medicine, Cairo University, and the Cancer Institute of New Jersey, UMDNJ/RWJMS
Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EGY-SCI-1
Record Dates: First submitted 2008-12-31; First posted 2009-01-05 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2009-01

CONDITIONS: Chronic Spinal Cord Injury
Keywords: Spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BM transplant with physiotherapy (Experimental): Autologous BM transplant
  Interventions: Procedure: Autologous bone marrow transplant; Procedure: Physical therapy
- Physiotherapy only (Active Comparator): conventional physical therapy for chronic spinal cord injury.
  Interventions: Procedure: Physical therapy

INTERVENTIONS:
Procedure: Autologous bone marrow transplant
  Arms: BM transplant with physiotherapy
Procedure: Physical therapy

SUMMARY:
This study is designed to assess the safety of autologous bone marrow derived cell transplant in chronic spinal cord injury patients. The hypothesis is that the availability of bone marrow derived mesenchymal stem cells at the sites of injury promote neuronal regeneration.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic spinal cord injury
* No concomitant systemic disease
* No progress on physiotherapy for at least 6 months
* Duration of injury from 10 months to 3 years

Exclusion Criteria:

* Non-traumatic spinal cord injury whether transverse myelitis or demyelination
* Concomitant systemic disease
* Progress can be observed on physiotherapy
* Acute injury or duration of injury less than 10 months

Ages: 10 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2005-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety of autologous BM transplant measured by absence of neuronal changes, infections or increased intracranial tension, and monitoring for any abnormal growth or tumor formation by MRI. | 18 months

SECONDARY OUTCOMES:
Efficacy of BM cell transplant in improving neurological functions in patients with chronic SCI. Improvement in motor, sensory and sphincteric functions, and quality of life using ASIA scores and MRI. | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University School of Medicine, Cairo, Egypt

REFERENCES:
- [Derived] El-Kheir WA, Gabr H, Awad MR, Ghannam O, Barakat Y, Farghali HA, El Maadawi ZM, Ewes I, Sabaawy HE. Autologous bone marrow-derived cell therapy combined with physical therapy induces functional improvement in chronic spinal cord injury patients. Cell Transplant. 2014 Apr;23(6):729-45. doi: 10.3727/096368913X664540. Epub 2013 Feb 26. PMID 23452836